CLINICAL TRIAL: NCT05017662
Title: A Multicentre Surveillance Study to Evaluate the Long-term Safety in Participants Who Have Been Previously Treated With 177Lu-IPN01072 in an Ipsen-sponsored Clinical Study
Brief Title: A Long-term Safety Surveillance Study in Participants Previously Treated With 177Lu-IPN01072
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariceum Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D-FR-01072-004; 2024-515071-35-00 (EU CTIS Number)
Record Dates: First submitted 2021-08-06; First posted 2021-08-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Data collection (Other)
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Participants will have surveillance visits every 3 months up to 5 years after their first dose of 177Lu-IPN01072 in Study OPS-C-001.

SUMMARY:
The purpose of the protocol is to evaluate the long-term safety of medicine 177Lu-satoreotide tetraxetan (also known as 177Lu-IPN01072 or 177Lu-OPS201) for patients who have previously received 177Lu-satoreotide tetraxetan in the clinical study OPS-C-001 / D-FR-01072-001.

DETAILED DESCRIPTION:
The study qualifies as interventional not because of the use of an investigational product, but because the imposed specific data collection includes assessments/blood collection and on-site visits not necessarily part of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of giving signed informed consent
* Participant must have received at least one infusion of 177Lu-IPN01072 in Study OPS-C-001

Exclusion Criteria:

- There are no exclusion criteria in this safety surveillance study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with second primary haematological and non-haematological malignancies. | During the whole study period (approximately 5 years).

SECONDARY OUTCOMES:
Proportion of treatment-related adverse events of any grade. | During the whole study period (approximately 5 years).
  Adverse events assessed according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE Version 5.0), including any treatment-related serious adverse events, as assessed by the investigators.
Changes over time in laboratory tests (haematology) | During the whole study period (approximately 5 years).
  Laboratory parameters (Platelet count, Haemoglobin and White Blood Cells count with differential) will be graded according to the NCI-CTCAE Version 5.0.
Changes over time in laboratory tests (biochemistry) | During the whole study period (approximately 5 years).
  Laboratory parameters (Creatinine) will be graded according to the NCI-CTCAE Version 5.0.
Overall survival defined as the time from the first dose of 177Lu-IPN01072 until death from any cause. | During the whole study period (approximately 5 years).

CONTACTS AND LOCATIONS:
Overall Officials: Ariceum Chief Medical Officer, Study Director — Ariceum
Locations (7):
- Australia (2):
  - Peter Maccallum Cancer Center, Melbourne
  - Ramsay Hollywood Private Hospital, Perth
- Medical University of Vienna, Vienna, Austria
- Aarhus University Hospital, Aarhus, Denmark
- Hôtel Dieu de Nantes, Nantes, France
- University Hospital Basel, Basel, Switzerland
- Royal Free Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes